CLINICAL TRIAL: NCT05206786
Title: Effectiveness of a Specific Strength Program of the Gluteus Maximus Muscle to Improve Dynamic Postural Control in Female Basketball Players
Brief Title: A Gluteus Maximus Strength Exercise Effectiveness for Improving Dynamic Postural Control in Female Basketball Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, Alexander Achalandabaso, Principal Investigator, University of Jaén
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEIM/2021/6/130
Record Dates: First submitted 2022-01-06; First posted 2022-01-25 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-05

CONDITIONS: Basketball
Keywords: Dynamic Postural Control; Gluteus Maximus; Lower limb; Injury prevention

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group. Conventional preventive work out (Experimental)
  Interventions: Other: Conventional preventive work out
- Intervention group. Gluteus maximus strengthening specific program (Experimental)
  Interventions: Other: Conventional preventive work out; Other: Gluteus maximus strengthening specific program

INTERVENTIONS:
Other: Conventional preventive work out — Female players in the control group will carry out a conventional preventive work that is organised in 3 training days per week. First training session includes preventive strength and proprioception exercises. Junior and senior teams (above 16 years old) will also do plyometrics exercises. In the second training session, players will do preventive strength exercises with an increased load compared to the previous session and proprioception exercises. Junior and senior players will also do anaerobic work. In the third session, players will perform reaction speed exercises.
Other: Gluteus maximus strengthening specific program — Female players will carry out a gluteus maximus strengthening work out in addition to the control group programme. Of the following four exercises, the first and the third ones will be done on the first training session and the second and the fourth exercises will be done on the second one. Dosage will be 2 sets of 10 repetitions for each leg.
  1. Clam Shell: Lateral decubitus with the knees and hips bend, the working leg placed on top of the other. Separate this knee while feet stay in contact.
  2. Unilateral gluteal bridge: Supine decubitus with one foot flat on the floor and bent knee. This leg pushes the ground with the foot until the pelvis is lifted while the other leg remains straight.
  3. Quadruped hip extension with knee extension : Quadruped on forearms. Straighten the hip by bringing the whole leg up and back with knee extension.
  4. Quadruped hip extension with bent knee: Performed as the previous one, but during this one, the knee of the working leg is bent at 90º.
  Arms: Intervention group. Gluteus maximus strengthening specific program

SUMMARY:
The study will be carried out at the Faculty of Nursing and Physiotherapy of the University of Alcalá. The study has been approved by the Animal Research and Experimentation Ethics Committee of the University of Alcalá. A total of 92 female basketball players aged between 12 and 25 will be selected and randomized in two different groups.

The control group will carry out a conventional preventive work out and the experimental group will carry out a specific strengthening program for the gluteus maximus in addition to the conventional preventive exercises.

The treatment will take place during the basketball club season and will last 4 months, from January to April 2022.

The objective is to evaluate the effectiveness of the inclusion of a specific gluteus maximus strength program in the conventional preventive work to improve the dynamic stability and to reduce the injury rate and pain in female basketball players.

ELIGIBILITY:
Inclusion Criteria:

* Female basketball players belonging to a sports club.
* Female basketball players between 12 and 25 years old.

Exclusion Criteria:

* Acute lower limb injuries at the start of the study.
* Surgery on the lower limb in the previous year.
* Injuries or diseases that prevent the correct performance of the evaluation tests.

Ages: 12 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 92 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Dynamic stability change assessed by a modified version of the Star Excursion Balance Test (SEBT). For this, Octobo-Balance device will be used. | Baseline and 4 months later
  Five lower limb excursion directions are going to be analysed: anterior (SEBT-A), medial (SEBT-M), posterior (SEBT-P), posteromedial (SEBT-PM) and posterolateral (SEBT-PL), with all these excursion directions and the legs' length of each player we will calculate the sum of them. The device system consists of an extending measuring tape magnetized to an octagon-shaped platform which allows to measure the different directions. There is a marked point in the middle of the octagon where players must put one of their feet properly and push the measuring tape with the other one. Players will have to go as far as possible in each direction without touching de floor or lifting the foot that it's set on the octagon. There will be three attempts in all the excursion directions, and it will be done for each leg.

SECONDARY OUTCOMES:
Change in the rate of lower limb injuries measured with a Daily Injury Report | Daily from baseline until the end of the research study 4 months later
  Lower limb injuries occurrence will be recorded on a daily basis. For this purpose, one person in charge of each team, under the supervision of the researchers, will fill in an injury report. This report will include basic information about the injury, so as the location, the side of the body, the type and the mechanism of the injury and the time of injury, as well as the happening and duration of a sick leave.
Pain change measured with the Visual Analogue Scale | Baseline and 4 months later
  Players will be asked to rate from 0 to 10 their general pain and their specific pain in: ankle, knee, hip and low back.
Vertical Jump Height using the app MyJump2 | Baseline and 4 months later
  Vertical jump is calculated analysing it on a recorded video with the help of this app. It is necessary to select manually the take-off frame and landing frame. Videos will be recorded by the researchers in the frontal plane in the same position and distance from the jumping player. Participants will be taught to perform a correct vertical jump, starting from a static position with knees and hips at 90º and the hands on the hips, as well as stretching the knees during the flight and landing. The objective is to achieve the maximum height with the jump. Total leg length (from anterior iliac spine to tiptoe in maximum plantar flexion) and height with flexed knees at 90º (measured vertically from floor to greater trochanter) will be measured to calculate the height of vertical jumps with the help of the app.
Dynamic knee valgus measured with the programme Kinovea | Baseline and 4 months later
  Players will be recorded from the frontal plane and in the same position for each player. Players shall perform three jumps in a row. Afterwards, with the Kinovea programme, the moment in which the highest knee valgus is produced in the landing of the different jumps will be analysed.
Treatment adherence through an exercise tracking diary | Weekly from baseline until the end of the research study 4 months later
  Players will be required to fill in a sheet in which they will be requested for whether or not they have done the corresponding exercises during the week.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Sánchez, Principal Investigator — University of Alcalá, Madrid, Spain
Locations (1):
- Sandra Sánchez, Alcalá de Henares, Madrid, Spain